CLINICAL TRIAL: NCT04832256
Title: Effects of Different Fresh Gas Flows on Carboxyhemoglobin Levels: Noninvasive Carbon Monoxide Monitoring
Brief Title: Effects of Different Fresh Gas Flows on Carboxyhemoglobin Levels
Status: Completed | Type: Observational
Sponsor: Zonguldak Bulent Ecevit University (Other)
Responsible Party: Principal Investigator, Bengü Gülhan Aydin, Associate Professor Doctor, Zonguldak Bulent Ecevit University
Other Study IDs: 2015-67-07/07
Record Dates: First submitted 2021-03-30; First posted 2021-04-05 (Actual); Last update posted 2022-05-03 (Actual); Status verified 2022-05

CONDITIONS: Fresh Flow; Carboxyhemoglobinemia
Keywords: Low flow anesthesia; Non-invasive carboxyhemoglobinemia monitoring; Smoking
MeSH Terms: conditions — Smoking

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- High Flow anesthesia: administered 4 L/min fresh gas flow during general anesthesia
  Interventions: Device: Radical-7 Pulse CO-Oximeter
- Low Flow Anesthesia: administered 1 L/min fresh gas flow during general anesthesia
  Interventions: Device: Radical-7 Pulse CO-Oximeter

INTERVENTIONS:
Device: Radical-7 Pulse CO-Oximeter — COHb measurement monitoring from finger pulp with a non-invasive measurement device called Masimo Radical-7 Pulse co-oximeter (Masimo Corporation, Irvine, USA)

SUMMARY:
To observe the effect of different fresh flows (1 L / min and 4 L / min) on the carboxyhemoglobin level non-invasively and continuous measurement and to determine the contribution of smoking to the intraoperative carbon monoxide accumulation.

ELIGIBILITY:
Inclusion Criteria:

* ASA I-II
* Undergo 2-4 hours of elective surgery

Exclusion Criteria:

* Cardiovascular disease
* diabetes mellitus
* kidney, liver failure
* chronic obstructive pulmonary disease
* patients with opioid sensitivity
* morbidly obese
* personal or family history of malignant hyperthermia
* history of prolonged recovery from anesthesia
* alcohol addicted
* pregnant and breastfeeding women patients allergic to study drugs

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: A total of 64 patients in ASA I-II risk group, aged 18-65, undergoing 2-4 hours of elective surgery
Sampling Method: Probability Sample
Enrollment: 64 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2019-06-01 (Actual)

PRIMARY OUTCOMES:
effects of different fresh gas flows on carboxyhemoglobin levels | during surgery
  To observe the effect of different fresh flows (1 L / min and 4 L / min) on the carboxyhemoglobin level by non-invasive and continuous measurement.

SECONDARY OUTCOMES:
effects of smoking on carbon monoxide accumulation. | during surgery
  to determine the contribution of smoking to intraoperative carbon monoxide accumulation.

CONTACTS AND LOCATIONS:
Locations (1):
- Zonguldak Bülent Ecevit University Medicine Faculty, Zonguldak, Kozlu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Koksal BG, Kucukosman G, Ozcan P, Baytar C, Bollucuoglu K, Okyay RD, Ayoglu H. Effects of different fresh gas flows on carboxyhemoglobin levels: non-invasive carbon monoxide monitoring: A randomized clinical trial. Saudi Med J. 2022 Aug;43(8):891-898. doi: 10.15537/smj.2022.43.8.20220424. PMID 35964947